CLINICAL TRIAL: NCT04480424
Title: A Multicenter, Randomized, Open-label Parallel Group Pilot Study to Evaluate Safety and Efficacy of High Dose Intravenous Immune Globulin (IVIG) Plus Standard Medical Treatment (SMT) Versus SMT Alone in Subjects With COVID-19 Requiring Admission to the Intensive Care Unit
Brief Title: Study to Evaluate the Safety and Efficacy of High Dose Intravenous Immune Globulin (IVIG) Plus Standard Medical Treatment (SMT) Versus SMT Alone in Participants in Intensive Care Unit (ICU) With Coronavirus Disease (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC2007
Record Dates: First submitted 2020-07-20; First posted 2020-07-21 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Coronavirus Disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2; Coronavirus Infections; Coronaviridae Infections; Virus Diseases; Immunoglobulins; Antibodies; Gamma-globulins; Immunoglobulins, Intravenous; Immunologic Factors; Physiological Effects of Drugs
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Coronaviridae Infections; Virus Diseases | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GAMUNEX-C + Standard Medical Treatment (Experimental): Participants received 2 grams per kilogram (g/kg) of GAMUNEX-C, which was capped to a maximum of 160 g infusion intravenously (IV) for participants weighing more than 80 kg on Day 1. The 2 g/kg net total dose was divided either into infusions of 500 mg/kg body weight over 4 days or 400 mg/kg body weight over 5 days as per investigator's decision. Participants received standard of care interventions as per Principal Investigator's discretion from Day 1 up to Day 29.
  Interventions: Biological: GAMUNEX-C; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Participants received all standard of care interventions required as per Principal Investigator's discretion throughout the participant's hospitalization, from Day 1 to Day 29.
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: GAMUNEX-C — Intravenous Immune Globulin (Human), 10% Caprylate/Chromatography Purified.
  Other Names: IGIV-C
  Arms: GAMUNEX-C + Standard Medical Treatment
Drug: Standard Medical Treatment — SMT per local policies or guidelines.

SUMMARY:
The purpose of the study is to determine if a high dose of Intravenous Immune Globulin (IVIG) plus Standard Medical Treatment (SMT) can reduce all-cause mortality versus SMT alone in hospitalized participants with COVID-19 requiring admission to the ICU through Day 29.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female subjects of ≥ 18 years of age at time of Screening who are being treated in the ICU for COVID-19 for not longer than 48 hours or for whom a decision has been made that COVID-19 disease severity warrants ICU admission.
* Has laboratory-confirmed novel coronavirus {SARS-CoV-2} infection as determined by qualitative polymerase chain reaction (PCR) (reverse transcriptase [RT]-PCR), or other United States Food and Drug Administration (FDA)-approved diagnostic assay for COVID-19 in any specimen during the current hospital admission prior to randomization.
* Illness (symptoms of COVID-19 of any duration requiring ICU level care), and the following:

  1. Radiographic infiltrates by imaging (chest X-Ray, computerized tomography (CT) scan, etc.), and
  2. Requiring mechanical ventilation and/or supplemental oxygen.
* Any one of the following related to COVID-19: i. Ferritin > 400 nanogram per milliliter (ng/mL), ii. Lactate dehydrogenase (LDH) > 300 units per liter (U/L), iii. D-Dimers > reference range, or iv. C-reactive protein (CRP) > 40 milligram per liter (mg/L).
* Subject provides informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Clinical evidence of any significant acute or chronic disease or pathophysiologic manifestations (eg, complications of COVID-19 standard medical treatments) that, in the opinion of the investigator, may place the subject at undue medical risk.
* The subject has had a known (documented) serious anaphylactic reaction to blood, any blood-derived or plasma product or a past history of any hypersensitivity reactions to commercial immunoglobulin.
* A medical condition in which the infusion of additional fluid is contraindicated.
* Shock that is unresponsive to fluid challenge and/or multiple vasopressors and accompanied by multiorgan failure considered by the Principal Investigator not able to be reversed.
* Subjects with known (documented) thrombotic complications to polyclonal IVIG therapy in the past.
* Subjects with current or prior myocardial infarction, stroke, deep vein thrombosis, or thromboembolic event (within the past 12 months) or who have a history of thromboembolic events of unknown etiology.
* Subjects with limitations of therapeutic effort.
* Female subjects who are pregnant or of child-bearing potential with a positive test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at Screening/Baseline.
* Subjects participating in another interventional clinical trial with investigational medical product or device.
* Known history of prothrombin gene mutation 20210, homozygous Factor V Leiden mutations, antithrombin III deficiency, protein C deficiency, protein S deficiency or antiphospholipid syndrome.
* Presence of malignancy (either new diagnosis of malignancy or known residual disease) within the past 12 months.
* Creatinine at Screening is ≥ 4 mg/dL (or subject is dependent on dialysis/renal replacement therapy).
* Known Immunoglobulin A (IgA) deficiency with anti-IgA serum antibodies.
* Uncontrolled hypertension at the time of Screening (systolic blood pressure > 200 mm Hg) or refractory severe hypotension with sustained systolic blood pressure < 90 mm Hg unresponsive to vasopressors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (18):
- United States (18):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Southern California Research Center, Coronado, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Via Christi Research, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - McLaren Flint, Flint, Michigan
  - McLaren Health Care-Macomb, Mount Clemens, Michigan
  - McLaren Health Care Oakland, Pontiac, Michigan
  - CHI Health, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - CHRISTUS Health, Tyler, Texas
  - MultiCare Deaconess Hospital, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 18 study centers in the United States. The study was conducted from 17 September 2020 to 25 October 2021.
Pre-assignment Details: Participants with Coronavirus Disease 2019 (COVID-19) were randomized in 1:1 ratio to receive Standard Medical Treatment (SMT) or SMT plus a net total dose of Gamunex-C of 2 grams per kilogram (g/kg) (body weight) administered in divided doses over 4 to 5 consecutive days at the Principal Investigator's discretion. Maximum dose was capped at 160 g.
Period: Overall Study
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Started | 50 | 50
Completed | 28 | 24
Not Completed | 22 | 26
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 14 | 16
Not completed — Reason not Specified | 5 | 5

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 55.5 [25 to 83] | 59.5 [26 to 79] | 57.5 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 24 | 27 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed is number of participants with data available for Ethnicity.
  Participants
    number analyzed (Participants) | 47 | 40 | 87
    Hispanic or Latino | 9 | 7 | 16
    Not Hispanic or Latino | 38 | 33 | 71
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 30 | 31 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Mortality Rate Through Day 29
Description: All-cause mortality rate is percentage of participants in each treatment group who experienced mortality up to Day 29.
Time Frame: Up to Day 29
Population: The intent to treat (ITT) population included all participants who were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
Percentage of participants | 28.0 | 32.0
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.8275, Fisher Exact — p-value was calculated using Fisher's exact method with 5% level of significance to test the null hypothesis of no difference in mortality rate between the two treatment groups; Risk Difference = -4.0, 95% CI 2-sided [-22.3 to 14.5]

2. Secondary Outcome: Percentage of Participants With Actual Intensive Care Unit (ICU) Discharge Time
Description: Percentage of participants who were discharged from ICU were recorded. Time to actual ICU discharge was defined as duration of actual ICU stay from Day 1 through Day 29.
Time Frame: Up to Day 29
Population: The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
Percentage of participants | 64 [48.9 to 75.7] | 62 [46.8 to 74.0]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.8599, Gray's test — p-value was calculated using Gray's test for equality of the Cumulative Incidence Function (CIF) between treatment groups

3. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration (number of days) of ICU stay from post-randomization through Day 29 was calculated based on ICU admission and discharge (actual and medical equivalence) dates.
Time Frame: Up to Day 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
days | 11.22 [8.01 to 14.43] | 8.64 [5.43 to 11.85]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.2626, ANOVA — p-value was calculated using an Analysis of Variance (ANOVA) model, including the number of days on mechanical ventilation as a dependent variable and treatment group as a fixed effect; Least Square Mean (LSM) Difference = 2.58, 95% CI 2-sided [-1.96 to 7.12]

4. Secondary Outcome: Percentage of Participants With Actual Hospital Discharge Time
Description: Percentage of participants who were discharged from the hospital were recorded. Time to hospital discharge was defined as duration of hospitalization from Day 1 through Day 29.
Time Frame: Up to Day 29
Population: The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
Percentage of participants | 62 [46.8 to 74.0] | 56 [41.0 to 68.6]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.6854, Gray's test — p-value was calculated using Gray's test for equality of the CIF between treatment groups

5. Secondary Outcome: Duration of Any Oxygen Use From Day 1 Through Day 29
Description: Duration (number of days) of any oxygen use from Day 1 through Day 29 was calculated based on the start/stop dates.
Time Frame: Up to Day 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
days | 23.00 [20.31 to 25.69] | 23.02 [20.33 to 25.71]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.9917, ANOVA — 95% CI for difference in least square mean (LSM) between treatment groups and the associated p-value were calculated using an ANOVA model, including the number of days on oxygen as a dependent variable and treatment group as a fixed effect; LSM Difference = -0.02, 95% CI 2-sided [-3.82 to 3.78]

6. Secondary Outcome: Mean Change From Baseline in Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. Higher score indicated no severe illness. Mean change in Ordinal scale was evaluated by fitting a linear mixed-effects model for repeated measures (MMRM). The data is reported for average across all postbaseline.
Time Frame: Baseline up to Day 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
score on a scale | -0.12 [-0.36 to 0.13] | -0.17 [-0.42 to 0.08]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.7557, Kenward-Roger; p-value were calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom; LSM Difference = 0.05, 95% CI 2-sided [-0.29 to 0.40]

7. Secondary Outcome: Absolute Change From Baseline in Ordinal Scale at Day 29
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities. Higher score indicated no severe illness.
Time Frame: Baseline, Day 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
score on scale | 1.05 [0.72 to 1.38] | 0.65 [0.32 to 0.98]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.0922, Kenward-Roger — p-value were calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom; LSM Difference = 0.40, 95% CI 2-sided [-0.07 to 0.86]

8. Secondary Outcome: Percentage of Participants in Each Severity Category of the 7-Point Ordinal Scale
Description: The ordinal scale is a 7-point scale ranging from 1 to 7 used to measure clinical status based on the following points: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Time Frame: Days 15 and 29
Population: The ITT population included all participants who were randomized. Number analyzed are the number of participants with data available for analysis at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
percentage of participants
  Day 15, Death: number analyzed (Participants) | 44 | 44
  Day 15, Death | 18.2 | 27.3
  Day 15, Hospitalized, on invasive mechanical ventilation or ECMO: number analyzed (Participants) | 44 | 44
  Day 15, Hospitalized, on invasive mechanical ventilation or ECMO | 31.8 | 15.9
  Day 15, Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 44 | 44
  Day 15, Hospitalized, on non-invasive ventilation or high flow oxygen devices | 11.4 | 18.2
  Day 15, Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 44 | 44
  Day 15, Hospitalized, requiring supplemental oxygen | 18.2 | 15.9
  Day 15, Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 44 | 44
  Day 15, Hospitalized, not requiring supplemental oxygen | 0 | 0
  Day 15, Not hospitalized, limitation on activities: number analyzed (Participants) | 44 | 44
  Day 15, Not hospitalized, limitation on activities | 13.6 | 20.5
  Day 15, Not hospitalized, no limitations on activities: number analyzed (Participants) | 44 | 44
  Day 15, Not hospitalized, no limitations on activities | 6.8 | 2.3
  Day 29, Death: number analyzed (Participants) | 41 | 40
  Day 29, Death | 31.7 | 40.0
  Day 29, Hospitalized, on invasive mechanical ventilation or ECMO: number analyzed (Participants) | 41 | 40
  Day 29, Hospitalized, on invasive mechanical ventilation or ECMO | 14.6 | 10.0
  Day 29, Hospitalized, on non-invasive ventilation or high flow oxygen devices: number analyzed (Participants) | 41 | 40
  Day 29, Hospitalized, on non-invasive ventilation or high flow oxygen devices | 2.4 | 2.5
  Day 29, Hospitalized, requiring supplemental oxygen: number analyzed (Participants) | 41 | 40
  Day 29, Hospitalized, requiring supplemental oxygen | 4.9 | 12.5
  Day 29, Hospitalized, not requiring supplemental oxygen: number analyzed (Participants) | 41 | 40
  Day 29, Hospitalized, not requiring supplemental oxygen | 2.4 | 0
  Day 29, Not hospitalized, limitation on activities: number analyzed (Participants) | 41 | 40
  Day 29, Not hospitalized, limitation on activities | 24.4 | 22.5
  Day 29, Not hospitalized, no limitations on activities: number analyzed (Participants) | 41 | 40
  Day 29, Not hospitalized, no limitations on activities | 19.5 | 12.5

9. Secondary Outcome: Percentage of Participants Who Develop Acute Respiratory Distress Syndrome (ARDS)
Description: Acute Respiratory Distress Syndrome was defined based on Berlin criteria (chest imaging, origin of edema, oxygenation).
Time Frame: Days 1, 5, 15 and 29
Population: The ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
percentage of participants
  Day 1 | 94.0 | 96.0
  Day 5 | 93.9 | 94.0
  Day 15 | 79.4 | 61.3
  Day 29 | 28.0 | 33.3

10. Secondary Outcome: Percentage of Participants Who Develop ARDS Distributed by Severity
Description: ARDS was defined by Berlin's criteria as: 1) Timing is usually within 1 week of a known clinical insult or new or worsening respiratory symptoms 2) Chest imaging: bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules 3) Respiratory failure not fully explained by cardiac failure or fluid overload Need objective assessment (eg, echocardiography) to exclude hydrostatic edema if no risk factor present 4) Oxygenation: Mild 200 mm Hg < partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) ≤ 300 mm Hg with positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP) ≥ 5 cm H2Oc; Moderate 100 mm Hg < PaO2/FIO2 ≤ 200 mm Hg with PEEP ≥ 5 cm H2O; Severe PaO2/FIO2 ≤100 mm Hg with PEEP ≥ 5 cm H2O.
Time Frame: Days 1, 5, 15 and 29
Population: The ITT population is included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
percentage of participants
  Day 1: Mild | 4.0 | 4.0
  Day 1: Moderate | 50.0 | 58.0
  Day 1: Severe | 40.0 | 34.0
  Day 5: Mild | 18.4 | 24.0
  Day 5: Moderate | 42.9 | 48.0
  Day 5: Severe | 32.7 | 22.0
  Day 15: Mild | 41.2 | 9.7
  Day 15: Moderate | 14.7 | 35.5
  Day 15: Severe | 23.5 | 16.1
  Day 29: Mild | 4.0 | 23.8
  Day 29: Moderate | 12.0 | 4.8
  Day 29: Severe | 12.0 | 4.8

11. Secondary Outcome: Change From Baseline in Sequential Organ Failure Assessment (SOFA) Score at Day 5, Day 15, and Day 29
Description: SOFA score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. The score is calculated on admission and every 24 hours until discharge using the worst parameters measured during the prior 24 hours SOFA score ranges from 0 (no organ dysfunction) to 24 (highest possible score / organ dysfunction). Higher score indicated severe illness.
Time Frame: Days 5, 15, and 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
score on a scale
  Change from Baseline at Day 5 | 0.34 [-0.28 to 0.95] | -0.07 [-0.68 to 0.55]
  Change from Baseline at Day 15 | 0.20 [-1.14 to 1.55] | 0.30 [-1.22 to 1.82]
  Change from Baseline at Day 29 | -0.87 [-2.58 to 0.83] | -0.95 [-2.98 to 1.08]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.3611, LSM Difference — p-value was calculated using restricted maximum likelihood with the Kenward-Roger method for calculating the denominator degrees of freedom; Kenward-Roger = 0.40, 95% CI 2-sided [-0.47 to 1.28]
Statistical Analysis 2: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.9238, LSM Difference — [p-value comment as in outcome 11, analysis 1]; Kenward-Roger = -0.10, 95% CI 2-sided [-2.13 to 1.94]
Statistical Analysis 3: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.9541, LSM Difference — [p-value comment as in outcome 11, analysis 1]; Kenward-Roger = 0.08, 95% CI 2-sided [-2.58 to 2.73]

12. Secondary Outcome: Change From Baseline in National Early Warning Score (NEWS)
Description: NEWS is clinical scoring developed to improve detection of deterioration in ill participant. It is based on 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure (BP), pulse rate, level of consciousness, and temperature. A score of 0 and 2 was allocated to supplemental oxygen, 0 and 3 for level of consciousness and score of 0, 1, 2 and 3 for remaining parameters (i.e. respiration rate, oxygen saturation, systolic BP, pulse rate and temperature) where 0 = normal health condition to 3 = worst health condition; higher score indicated more severity. All scores were summed to get an aggregate score. Aggregate NEWS score ranged from 0 to 20, with higher scores meaning more severity/higher risk.
Time Frame: Baseline and Day 29
Population: The ITT population included all participants who were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
score on a scale | -2.56 [-3.56 to -1.57] | -2.62 [-3.71 to -1.54]
Statistical Analysis 1: Comparison: GAMUNEX-C + Standard Medical Treatment vs Standard Medical Treatment; Test type: Superiority; p = 0.9366, LSM Difference — [p-value comment as in outcome 11, analysis 1]; LSM Difference = 0.06, 95% CI 2-sided [-1.42 to 1.53]

13. Secondary Outcome: Percentage of Participants Achieving Clinical Response: NEWS ≤ 2 Maintained for 24 Hours
Description: Percentage of participants who achieved clinical response (i.e the NEWS score ≤2 maintained for 24 hours from Day 1 through Day 29) was estimated using the Kaplan-Meier method.
Time Frame: Day 29
Population: The ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
Number analyzed (Participants) | 50 | 50
percentage of participants | 32.9 [18.5 to 54.1] | 28.2 [14.8 to 49.5]

ADVERSE EVENTS:
Time Frame: From the start of the study up to Day 90
Arm/Group | GAMUNEX-C + Standard Medical Treatment | Standard Medical Treatment
All-Cause Mortality (participants affected / at risk) | 16/50 | 18/50
Serious Adverse Events (participants affected / at risk) | 27/50 | 23/50
Other Adverse Events (participants affected / at risk) | 42/50 | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GAMUNEX-C + Standard Medical Treatment (N=50) | Standard Medical Treatment (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 4 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Meningism (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Distributive shock (Vascular disorders) | 1 | 0
Hypoperfusion (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GAMUNEX-C + Standard Medical Treatment (N=50) | Standard Medical Treatment (N=50)
Anemia (Blood and lymphatic system disorders) | 6 | 6
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 5
Bradycardia (Cardiac disorders) | 4 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 5 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Eye disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 2 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Tachyphylaxis (General disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0
Herpes dermatitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia bacterial (Infections and infestations) | 4 | 1
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 1
Pneumonia serratia (Infections and infestations) | 0 | 1
Salpingitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Perineal injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 1 | 1
Blood creatinine decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood pH increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Body temperature decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 2 | 1
C-reactive protein increased (Investigations) | 1 | 1
Carbon dioxide increased (Investigations) | 1 | 0
Coombs direct test positive (Investigations) | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 2 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Heart rate abnormal (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 2 | 0
Occult blood positive (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Platelet count increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Respiratory rate increased (Investigations) | 4 | 2
Serum ferritin increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 8
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 3
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Intensive care unit delirium (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 1
Tracheostomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Distributive shock (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 11 | 10
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Microembolism (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Vasodilatation (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT04480424/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT04480424/SAP_001.pdf